CLINICAL TRIAL: NCT05191498
Title: Intratumoral Holmium Microspheres Brachytherapy for Patients With Pancreatic Cancer; a Single Center, Non-randomized, Feasibility Study in an Open Surgical Setting - the SLOTH1 Study
Brief Title: Intratumoral Holmium Microspheres Brachytherapy for Patients With Pancreatic Cancer
Acronym: SLOTH-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Quirem Medical B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL76311.091.20
Record Dates: First submitted 2022-01-02; First posted 2022-01-13 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2023-05

CONDITIONS: Pancreas Cancer
Keywords: Intratumoral therapy; Holmium microspheres
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study patients (Experimental): All patients receive intratumoral holmium microsphere injections ones, if surgery is suspended. Patient specific treamtent planning is performed for every individual patient.
  Interventions: Device: QuiremSpheres®

INTERVENTIONS:
Device: QuiremSpheres® — Intratumoral injection of QuiremSpheres® up to a dose of 150 Gy.

SUMMARY:
This is a feasibility study in which patients with pancreatic cancer are treated with intratumoral holmium microsphere injections.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male aged 18 years and over.
2. Diagnosis of primary (borderline) resectable pancreatic cancer by Dutch Pancreatic Cancer Group (DPCG) guidelines:

   i. 1o-90o contact between tumor and the superior mesenteric artery, celiac axis or common hepatic artery. Or; ii. 90o-270o contact between tumor and superior mesenteric vein or portal vein, without occlusion.

   iii. The discussion on resectability has to be made in consensus at multidisciplinary meetings/discussions and may overrule the above criteria (i, ii).
3. Patient is deemed eligible for surgical resection of the pancreatic cancer, however, during open surgery a more advanced disease than initially anticipated is found and resection is no longer feasible.
4. Life expectancy of 12 weeks or longer.
5. World Health Organisation (WHO) Performance status 0-1.
6. One or more measurable lesions of at least 10 mm in the longest diameter by spiral CT or MRI according to the Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 criteria.
7. Negative pregnancy test for women of childbearing potential.

Exclusion Criteria:

1. Radiation therapy within the last 4 weeks before the start of study therapy.
2. Calcifications in the pancreas or tumour that are highly expected to obstruct the needle tract
3. Any unresolved toxicity greater than National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (CTCAE version 4.0) grade 2 from previous anti-cancer therapy.
4. Leukocytes < 4.0 109/l and/or platelet count < 100 109/l.
5. Significant cardiac event (e.g. myocardial infarction, superior vena cava (SVC) syndrome, New York Heart Association (NYHA) classification of heart disease ≥2 within 3 months before entry, or presence of cardiac disease that in the opinion of the Investigator increases the risk of ventricular arrhythmia.
6. Patient is deemed ineligible for implantation of 166Ho by an expert panel (surgeon, nuclear medicine physician and researcher) due to tumour anatomy or nearby structures.
7. Pregnancy or breast feeding (women of child-bearing potential).
8. Patients suffering from psychic disorders that make a comprehensive judgement impossible, such as psychosis, hallucinations and/or depression.
9. Patients who are declared incompetent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2024-02-18 (Actual); Study Completion 2024-02-18 (Actual)

PRIMARY OUTCOMES:
Average tumour dose by SPECT imaging | At 1 week after intervention
  To establish the feasibility of intratumoral implantation of QuiremSpheres® by evaluating the average tumour absorbed dose in Gy calculated on SPECT.

SECONDARY OUTCOMES:
Microsphere distribution by MRI | At 1 week after intervention
  Microsphere distribution in analysed using MRI to evaluate tumour absorbed and non-target absorbed dose.
Microsphere distribution by CT | At 1 week after intervention
  Microsphere distribution in analysed using CT to evaluate tumour absorbed and non-target absorbed dose.
Number of treatment-related adverse events as assessed by CTCAE v4.0 | Up to 3 months after intervention
  Safety, expressed in Common Terminology Criteria for Adverse Events, grade 3 and higher, probably or definitely related to the implantation procedure or medical device implant is monitored up to 3 months after intervention.
Tumor response by RECIST 1.1 | At 3 months after intervention
  Tumor response to the intervention is evaluated according to the Response evaluation criteria in solid tumors (RECIST) version 1.1 after 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Nijsen, PhD, Principal Investigator — Associate professor
Locations (1):
- Radboud University Medical Centre, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided